CLINICAL TRIAL: NCT01711242
Title: Phase II Randomized Trial of Adjuvant XELOX Chemotherapy and XELOX With Concurrent Capecitabine and Radiotherapy for Gastric Adenocarcinoma With D2 Dissection
Brief Title: Trial of Adjuvant XELOX Chemotherapy and Concurrent Capecitabine and Radiotherapy for Resected Gastric Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: xie congying (Other)
Responsible Party: Sponsor-Investigator, xie congying, Director, Wenzhou Medical University
Organization: Wenzhou Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: WZMC-12068
Record Dates: First submitted 2012-10-14; First posted 2012-10-22 (Estimated); Last update posted 2022-05-05 (Actual); Status verified 2022-04

CONDITIONS: Gastric Cancer
Keywords: gastric cancer; radiotherapy; postoperative therapy; chemotherapy
MeSH Terms: conditions — Stomach Neoplasms | interventions — Capecitabine; Oxaliplatin; Radiotherapy

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- capecitabine/Oxaliplatin/radiotherapy (Experimental): sequence chemoradiotherapy following radical resection
  sequence chemoradiotherapy two cycles of XELOX + concurrent chemoradiotherapy + two cycles of XELOX.
  Postoperative radiotherapy regimen: Radiotherapy consisted of 4500 centigray of radiation at 180 centigray per day, five days per week for five weeks, to the tumor bed, to the margins of resection or the stoma, to the regional nodes. Protection of spinal cord, heart, liver and kidney should be considered.
  Concurrent chemotherapy regimen: capecitabine 825 mg/m² twice daily Postoperative chemotherapy regimen: see arm 2
  Interventions: Drug: Capecitabine; Drug: Oxaliplatin; Radiation: Radiotherapy
- capecitabine/Oxaliplatin (Active Comparator): chemotherapy alone following radical resection
  Drug: chemotherapy alone following radical resection Postoperative chemotherapy regimen: The XELOX regimen was administrated: Oxaliplatin, 130mg/m2/day on day1, i.v. 2h; Capecitabine 1000mg/m²/day twice daily d1-14; every 21 days repeated, for 4 cycles.
  Interventions: Drug: Capecitabine; Drug: Oxaliplatin

INTERVENTIONS:
Drug: Capecitabine
Drug: Oxaliplatin
Radiation: Radiotherapy
  Arms: capecitabine/Oxaliplatin/radiotherapy

SUMMARY:
The objective of the trial is to compare disease-free survival between adjuvant XELOX alone vs XELOX with concurrent capecitabine and radiotherapy in curatively resected gastric cancer patients with D2 dissection.

DETAILED DESCRIPTION:
Gastric cancer is one of the most common malignancies in China. Complete surgical resection is the only potentially curative therapy available to patients with gastric cancer. However, the overall survival results remain unsatisfactory. The main factor accounting for high mortality rate is the relapse after surgical resection. During the past few decades, the principle of combined modality treatment has been developed and applied in gastric cancer. Radiation therapy plus concurrent chemotherapy had demonstrated to be able to achieve a significant improvement in overall and disease-free survival according to Intergroup Trial 0116/Southwest Oncology Group 9008. Nevertheless, the result from Intergroup Trial 0116 study had been challenged by the fact that the surgical treatment applied in the trial was gastrectomy with limited lymph node dissection (D0 or D1) in 90% of cases. Therefore, it is debatable whether adjuvant chemoradiation therapy can confer survival benefit in patients with extensive lymph node dissection. In ARTIST study, the addition of concurrent capecitabine and radiotherapy to capecitabine and cisplatin chemotherapy did not significantly reduce recurrence after curative resection and D2 lymph node dissection in gastric cancer. In subgroup analysis of patients with positive pathologic lymphnodes, there was a statistically significant prolongation in disease-free survival in the concurrent treatment arm when compared with the chemotherapy alone arm. Furthermore, CLASSIC study showed that XELOX (oxaliplatin/capecitabine) combination given as adjuvant chemotherapy for stage II or III patients after D2 surgery could achieve a significant survival benefit. The standard treatment modality in gastric cancer after D2 dissection is still disputable. Thus, the assessment of the effect of adjuvant sequence chemoradiotherapy in D2 resected gastric cancer is essential.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven gastric cancer; ≥ D2 resection
* Stage T1-4, N+
* 18 ≤ age ≤ 75
* Eastern Cooperative Oncology Group 0-2
* No distant metastasis
* Adequate bone marrow functions (absolute neutrophil count≥ 1,500/ul, blood platelet≥ 100,000/ul, haemoglobin≥ 10g/dl)
* Adequate renal functions(serum creatinine ≤ 1.5mg/dl)
* Adequate liver functions (serum bilirubin ≤ 1.5mg/dl, aspartate aminotransferase/alanine aminotransferase ≤ 3 times(normal value)
* Written informed consent

Exclusion Criteria:

* Previous history of immunotherapy, chemotherapy, radiotherapy for gastric cancer;
* Active infection requiring antibiotics;
* Pregnant, lactating women;
* Psychiatric illness, epileptic disorders;
* Concurrent systemic illness not appropriate for chemotherapy;
* Resection margin (+);
* History of other malignancy within 5 years except for non-melanoma skin cancer, cervix in situ carcinoma;
* D0, D1 resection;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Actual)
Dates: Start 2012-01 (Actual); Primary Completion 2020-01 (Actual); Study Completion 2021-01 (Actual)

PRIMARY OUTCOMES:
disease free survival | 3-year

SECONDARY OUTCOMES:
5 year Overall Survival | 5 years

OTHER OUTCOMES:
Health-related quality of life | five years after enrollment
  assessed by the Functional Assessment of Cancer Therapy-Esophageal (FACT-E)
Number of participants with adverse events as a measure of safety and tolerability | during treatment
  assessed by NCI Common Terminology Criteria v3.0

CONTACTS AND LOCATIONS:
Overall Officials: congying xie, MD, Principal Investigator — First Affiliated Hospital of Wenzhou Medical University; xiaolei chen, MD, Principal Investigator — First Affiliated Hospital of Wenzhou Medical University
Locations (1):
- The First Affiliated Hospital of Wenzhou Medical College, Wenzhou, Zhejiang, China